CLINICAL TRIAL: NCT00445250
Title: Phase 2 Study of the Role of Calcipotriol as Radioprotector of Skin in Women Receiving Radiotherapy Treatment to the Breast.
Brief Title: The Role of Calcipotriol as Radioprotector of Skin
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 004253
Record Dates: First submitted 2007-03-07; First posted 2007-03-08 (Estimated); Last update posted 2007-03-08 (Estimated); Status verified 2007-01

CONDITIONS: Radiodermatitis
Keywords: Calcipotriol; Breast; Cancer; Radiotherapy; Radiodermatitis in Breast Cancer
MeSH Terms: conditions — Radiodermatitis; Neoplasms | interventions — calcipotriene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Calcipotriol

SUMMARY:
Examining the hypothesis that protecting keratinocytes by calcipotriol can prevent in-vivo cutaneous side effect in patients receiving radiotherapy to the breast.

To check the connection between the skin effect of radiotherapy and different parameters including diseases such as diabetes and lupus, use of medications, allergies, weight, habits, size of the irradiated breast, previous chemotherapy treatment and exposure to sunlight.

DETAILED DESCRIPTION:
STUDY PROTOCOL

Fifty women diagnosed with breast cancer planned to receive adjuvant radiotherapy, will participate in the study. About 15 minutes after receiving the daily radiation dose fraction, a cream containing an active vitamin D analogue will be applied to half of the breast with inspection of a nurse. The other half of the breast will have a standard cream applied . During the days that radiotherapy is not administered the standard cream will be applied to both halves of the breast in a case of strong reaction to radiotherapy (e.g. strong erythema, painful tenderness etc.)The adverse skin effects will be assessed according to the following criteria:

1. . an assessment by a physician and a nurse according to the RTOG score (6).

   As follows:

   Grade 0 - no reaction. Grade 1 - light erythema dry peeling, decrease in sweat production. Grade 3 - extensive moist peeling, pitting edema. Grade 4 - ulcers, bleeding and necrosis.
2. . A questionnaire to each patient regarding the efficacy and safety of the cream.
3. . Number of interruption of radiotherapy treatment. The assessment will be done each week during radiotherapy treatment and weekly for three weeks following the completion of radiotherapy treatment.

Safety report will be sent to the local independent ethics committee after the examination of the first ten patients.

The protective effect of the cream containing calcipotriol will be compared to the standard treatment and analyzed statistically using the parameters mention above. The relation between the background disease, medications, allergies, weight, habits, size of the irradiated breast, sun exposure, previous chemotherapy treatment and exposure to sunlight and the skin reaction will be evaluated.

INCLUSION CRITERIA

1. . Age ranging from 18 to 75.
2. . Confirmed histological diagnosis of Breast cancer.
3. . Radiotherapy treatment to the breast following lumpectomy.

EXCLUSION CRITERIA

1. . Scleroderma.
2. . An extremely large breast. Interfiled above 25 cm.
3. . Prior radiotherapy to the same breast, radiotherapy to the contra lateral breast is not a contraindication.
4. . Mastectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ranging from 18 to 75.
2. Confirmed histological diagnosis of Breast cancer.
3. Radiotherapy treatment to the breast following lumpectomy.

Exclusion Criteria:

1. Scleroderma.
2. An extremely large breast. Interfiled above 25 cm.
3. Prior radiotherapy to the same breast, radiotherapy to the contra lateral breast is not a contraindication.
4. Mastectomy.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50

PRIMARY OUTCOMES:
Prevention of radiodermatitis

SECONDARY OUTCOMES:
Side effects of Calcipotriol

CONTACTS AND LOCATIONS:
Overall Officials: Eyal Fenig, M.D., Principal Investigator — Rabin Medical Center
Locations (1):
- Rabin Medical Center, Petach Tiqva, Israel